CLINICAL TRIAL: NCT04783402
Title: A Telehealth-based Cognitive-adaptive Training for Women With Breast Cancer in Risk to Suffer Cancer and Chemotherapy-related Cognitive Impairment: a Randomized Controlled Trial.
Brief Title: Telehealth Program to Prevent Cancer and Chemotherapy-related Cognitive Impairment.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Lydia Mª Martín-Martín, Lecturer, PhD researcher and investigator, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: e-OTCAT20
Record Dates: First submitted 2021-02-21; First posted 2021-03-05 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Breast Neoplasms
Keywords: Chemotherapy; Occupational Therapy; Quality of Life; Cognitive Impairment; Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms; Cognitive Dysfunction | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- e-OTCAT (Experimental): The experimental group will receive the e-OTCAT program that consists of a 12-week videoconference-based occupational therapy intervention at the same time women with breast cancer receive chemotherapy.
  Interventions: Other: e-OTCAT program
- Control Group (Other): At the beginning of chemotherapy, the participants allocated to the control group will only receive an educational handbook containing information about most frequent side-effects of cancer and cancer treatments, plus standard care for these patients.
  Interventions: Other: Educational handbook and standard care

INTERVENTIONS:
Other: e-OTCAT program — The e-OTCAT program consists of a combination of cognitive training in terms of attention, memory and processing speed; and adaptive training based on metacognition and cognitive-behavioral strategies (psycho-education, relaxation techniques training, stress management, energy conservation techniques, time management, etc.).
  This program also includes homework exercises consisting of a handbook of paper-and-pencil exercises, a cognitive training mobile app, and the practice of strategies seen in adaptive training sessions.
  Arms: e-OTCAT
Other: Educational handbook and standard care — At the beginning of chemotherapy, the participants will receive an educational handbook containing information about most frequent side-effects of cancer and cancer treatments, plus standard care.
  Arms: Control Group

SUMMARY:
The present randomized controlled trial has the main objective to study the effects of a videoconferenced occupational therapy program in preventing cancer and chemotherapy-related cognitive impairment and other health outcomes, as well as in improving quality of live and occupational performance of women undergoing chemotherapy for breast cancer.

DETAILED DESCRIPTION:
The chemotherapy-related cognitive impairment (also called chemobrain) has a great incidence among breast cancer population. However, the knowledge about effective interventions of supportive care is still inconsistent. Furthermore, the majority of programs targeted to this problem has been applied in survivorship, while the onset of cognitive impairment and the decline in quality of life occur during medical treatments. In this line, actual evidence suggests testing the effectiveness of interventions in a preventive setting in patients with breast cancer scheduled to receive neurotoxic chemotherapy. In addition, telehealth approaches have become a promising practice and increasingly more frequent among healthcare disciplines.

Our objective is to study the effects of a videoconferenced cognitive training in combination with cognitive-behavioral strategies to prevent or mitigate the cancer- and chemotherapy-related cognitive impairment in women with breast cancer who undergo this treatment, as well as to improve quality of life and allow an optimal adaptation to the occupational needs derived from medical treatment.

This study will use a two-arm, single blinded randomized clinical trial design. Eligible women will be randomized to one of the following groups: the experimental group that will receive the e-OTCAT program (12 weeks), or the control group that will receive and educational handbook and standard care. The study outcomes will be assessed after intervention and at 6-month follow-up post-randomization.

This study may contribute the need to include disciplines such as occupational therapy in the supportive care of cancer patients during the active phase of the disease, as well as the potential advantages provided by a telehealth approach related to economic, temporal and geographical barriers.

ELIGIBILITY:
Inclusion Criteria:

* Female with breast cancer who are going to start chemotherapy
* Stage I-III breast cancer
* No evidence of disease at time of screening
* Must be able to speak, read and write Spanish well to complete written and verbal assessment, neurocognitive tests and study tasks
* Must have basic phone skills

Exclusion Criteria:

* History of neurological disorder with cognitive symptoms (i.e., Parkinson's disease, Alzheimer disease, seizure disorder, multiple sclerosis, etc.)
* History of psychiatric disorder such as mental retardation, bipolar disorder, schizophrenia, etc.
* History of traumatic brain injury with ≥ 30' of consciousness or cognitive sequelae as per self-report or as documented in the medical record
* Prior history of cancer or secondary diagnosis of cancer
* Prior history of chemotherapy
* A hearing or visual deficit

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2020-10-31 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Subjective cognitive Function: | Participants will be followed over 6 months
  The primary outcome will be assessed with the Functional Assessment of Cancer Therapy-Cognitive Function (FACT-Cog) will be used to assess the subjective cognitive functioning.

SECONDARY OUTCOMES:
Objective Cognitive Function: Attention | Participants will be followed over 6 months
  The Trail Making Test (A and B parts) will be used to assess speed for attention, sequencing, mental flexibility, visual search and motion function. Time spent in each part is noted. Lower results (less time) indicate better test performance.
Objective Cognitive Function: Verbal Memory | Participants will be followed over 6 months
  The Rey Auditory Verbal Learning Test will be used to assess verbal memory and learning. A greater number of remembered words indicate better performance.
Objective Cognitive Function: Working Memory and Processing Speed | Participants will be followed over 6 months
  Wechsler Adult Intelligence Scale (WAIS-IV) will be used to assess working memory and processing speed. We will use the following tests: digit span, arithmetic, symbol search and coding. Higher scores in each test indicate a better cognitive performance.
Psychological status | Participants will be followed over 6 months
  The Hospital Anxiety and Depression Scale (HADS) will be used to assess levels of anxiety and depression. In the HADS subscales (anxiety and depression), scores ranging from 0 to 21. Scores between 8-10 indicate suspicious case of anxiety or depression, and scores higher than 11 are likely cases of anxiety or depression.
Cancer-Related Fatigue | Participants will be followed over 6 months.
  The Piper Fatigue Scale-Revised (PFS-R) will be used to assess the presence of cancer-related fatigue. Items are grouped into four dimensions (behavioral, cognitive, sensorial and affective) obtaining a global score. Higher results indicate a higher level of fatigue.
Quality of Sleep | Participants will be followed over 6 months.
  The Pittsburgh Sleep Quality Index (PSQI) will be used to assess the quality of sleep through the following dimensions: quality, latency, duration, efficiency, alterations, use of medication and daily dysfunction. A total score is obtained ranging from 0 to 21. Higher scores indicate a poor quality of sleep.
Occupational Performance | Participants will be followed over 6 months
  The Canadian Occupational Performance Measure (COPM) will be used to assess the self-perception of performance and satisfaction with activities of daily living.
Overall Quality of Life | Participants will be followed over 6 months
  The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 version 3.0 will be used to assess quality of life. The EORTC QLQ-C30 is composed of five functional scales (role, physical, cognitive, emotional and social), a global quality of life scale and nine symptom scales (fatigue, nausea and vomiting, pain, dyspnea, sleep disturbance, appetite loss, constipation, diarrhea and financial impact). Higher scores in the first two subscales indicate better function and quality of life, while higher scores in the symptom scales indicate a major impact of those symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Granada, Granada, Spain

REFERENCES:
- [Derived] Gonzalez-Santos A, Lopez-Garzon M, Sanchez-Salado C, Postigo-Martin P, Lozano-Lozano M, Galiano-Castillo N, Fernandez-Lao C, Castro-Martin E, Gallart-Aragon T, Legeren-Alvarez M, Gil-Gutierrez R, Martin-Martin L. A Telehealth-Based Cognitive-Adaptive Training (e-OTCAT) to Prevent Cancer and Chemotherapy-Related Cognitive Impairment in Women with Breast Cancer: Protocol for a Randomized Controlled Trial. Int J Environ Res Public Health. 2022 Jun 10;19(12):7147. doi: 10.3390/ijerph19127147. PMID 35742400